CLINICAL TRIAL: NCT07344987
Title: A Randomized Crossover Trial of Indoor Air Quality Improvement on Health in Patients With Interstitial Lung Disease
Brief Title: Effect of Indoor Air Quality Improvement on Health in Patients With Interstitial Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Hongbing Xu, Prof., Peking Union Medical College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CAMS-PUMC-IRM-IAQ-ILD-2025
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: ILD
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purifier (without Filter) Arm (Sham Comparator)
  Interventions: Behavioral: Purifier (without Filter) Arm
- Air Purifier (with Filter) Arm (Experimental)
  Interventions: Behavioral: Air Purifier (with Filter) Arm

INTERVENTIONS:
Behavioral: Air Purifier (with Filter) Arm — Place an air purifier with high-efficiency filters in the home, and turn it on for at least 18 hours every day.
  Arms: Air Purifier (with Filter) Arm
Behavioral: Purifier (without Filter) Arm — Place an air purifier without a filter in the home.
  Arms: Purifier (without Filter) Arm

SUMMARY:
Air pollution threatens the respiratory health of patients with interstitial lung disease (ILD). High-efficiency air purifiers, featuring easy operation and excellent particulate matter removal efficiency, have been shown in previous studies to potentially delay lung function deterioration and reduce acute exacerbation risk in respiratory disease patients. This randomized crossover study employs air purifiers to filter indoor gaseous pollutants, allergens, and other contaminants, aiming to alleviate respiratory irritation, improve daily life comfort, and enhance overall health status in ILD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with interstitial lung disease (ILD).
* Stable disease status, defined as no hospitalization due to acute exacerbation within the past month.

Exclusion Criteria:

* Patients with complications of severe organ failure (including heart, liver, or kidney failure), malignant tumors, or mental disorders.
* A history of respiratory tract infection within the past two weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Symptom Improvement-related Indicators (e.g., Improvement in Respiratory Symptom Score) | Baseline (before intervention), Week 2 (end of first phase), Week 6 (end of second phase)
  St. George's Respiratory Questionnaire (SGRQ):Score Range:Minimum score: 0 points;Maximum score: 100 points.A higher score indicates worse outcomes for the patient.
Pulmonary Function Indicators (e.g., Pulmonary Diffusing Capacity) | Baseline (before intervention), Week 2 (end of first phase), Week 6 (end of second phase)
Quality of Life Indicators (e.g., CAT Score) | Baseline (before intervention), Week 2 (end of first phase), Week 6 (end of second phase)
  COPD Assessment Test (CAT):It is a short, validated, patient-reported outcome (PRO) tool specifically designed to measure the impact of pulmonary disease on a patient's health status and daily life.Score Range:Minimum score: 0 points;Maximum score: 40 points.A higher score indicates worse health status and greater pulmonary disease-related burden for the patient.
Blood Sample Indicators (e.g., Concentration of Interleukin-8) | Baseline (before intervention), Week 2 (end of first phase), Week 6 (end of second phase)
  Assessment of Changes in Pulmonary Inflammation or Lung Injury Before and After Intervention Using Concentrations of Biomarkers Such as Interleukin-8

IPD SHARING:
Plan to Share IPD: No
1. The informed consent form signed by study participants does not include clauses authorizing the sharing of de-identified individual participant data (IPD) with external researchers. In accordance with the ethical approval requirements, no secondary use of IPD beyond the primary study objectives is permitted without explicit participant consent.
  2. The sample size of this study is relatively small, and the collected IPD has high heterogeneity due to individual differences in patient clinical characteristics and intervention responsiveness. Sharing such a limited dataset may not support robust secondary research findings, and could lead to misleading interpretations of the intervention effect on pulmonary inflammation.